CLINICAL TRIAL: NCT01926392
Title: A Prospective Randomized Trial Comparing Silver Sulfadiazine Cream to a Water-Soluble Poly-Antimicrobial Gel in Partial Thickness Burn Wounds
Brief Title: Comparison of a Water-soluble Topical Antimicrobial to Silver Sulfadiazine in Partial Thickness Burns
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 15603
Record Dates: First submitted 2013-08-17; First posted 2013-08-20 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: Burn
MeSH Terms: conditions — Burns | interventions — Silver Sulfadiazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- water-soluble therapy (Experimental): The patient acted as their own control and the experimental and comparison arms (water-soluble therapy and silver sulfadiazine) were alternated on a daily basis
  Interventions: Drug: water-soluble therapy; Drug: silver sulfadiazine
- silver sulfadiazine (Active Comparator): The patient acted as their own control and the experimental and comparison arms (water-soluble therapy and silver sulfadiazine) were alternated on a daily basis
  Interventions: Drug: water-soluble therapy; Drug: silver sulfadiazine

INTERVENTIONS:
Drug: water-soluble therapy — The patient acted as their own control and the experimental and comparison arms (water-soluble therapy and silver sulfadiazine) were alternated on a daily basis
Drug: silver sulfadiazine — The patient acted as their own control and the experimental and comparison arms (water-soluble therapy and silver sulfadiazine) were alternated on a daily basis

SUMMARY:
Partial thickness burns are a common, painful injury requiring a great deal of resources in their care. Silver sulfadizine is a commonly-used topical antimicrobial, but is difficult to remove due to its lipid base. We are comparing a water-based topical antimicrobial therapy to silver sulfadiazine and hypothesize that the water-based therapy is superior in terms of pain control and resources required to deliver care.

ELIGIBILITY:
Inclusion Criteria:

* adult inpatients with partial thickness burns

Exclusion Criteria:

* superficial or full thickness burns, facial burns, intubated or sedated, pediatric

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Pain level | 180 minutes
  Pain is assessed on a 0-10 point scale using both the patient's reported value and correlating with the value derived from nursing assessment using the visual analog scale. This is recorded at defined time points before, during, and after the dressing change

SECONDARY OUTCOMES:
time to perform dressing changes | up to 180 minutes
  The time to perform the dressing change in total and for various steps is recorded in minutes.

OTHER OUTCOMES:
narcotic medication administered | 180 minutes
  All narcotics given for premedication and during the dressing change will be converted to their morphine-equivalent and totaled

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Black, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States